CLINICAL TRIAL: NCT04555408
Title: Efficacy of Blue Light Treatment in Patients With Nonseasonal Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Mental Health Center, Jingan District (Other); Shanghai Mental Health Center, Yangpu District (Unknown); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019ZSQN44
Record Dates: First submitted 2020-09-15; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-07

CONDITIONS: Depression
Keywords: nonseasonal major depression disorder; light therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- blue light group (Active Comparator): The blue light will be applied five times a week for the first two weeks. For the next two weeks, this treatment will be applied three times a week.
  Interventions: Device: blue light
- bright light group (Active Comparator): The bright light will be applied five times a week for the first two weeks. For the next two weeks, this treatment will be applied three times a week.
  Interventions: Device: bright light
- dim light group (Placebo Comparator): The dim light will be applied five times a week for the first two weeks. For the next two weeks, this treatment will be applied three times a week.
  Interventions: Device: dim light

INTERVENTIONS:
Device: blue light — Patients receive exposure to 100lux blue light, which dominant wave-length is 468nm for 30 minutes in the morning.
  Arms: blue light group
Device: bright light — Patients receive exposure to 1000lux bright light, which dominant wave-length is 490nm for 30 minutes in the morning.
  Arms: bright light group
Device: dim light — Patients receive exposure to 100lux dim light, which dominant wave-length is 490nm for 30 minutes in the morning.
  Arms: dim light group

SUMMARY:
To compare the efficacy of blue light, bright light and dim light in the treatment of with nonseasonal major depression disorder(MDD) in adults.

DETAILED DESCRIPTION:
The current study aims to compare the efficacy of blue light, bright light and dim light in the treatment of with nonseasonal major depression disorder(MDD) in adults. 162 patients with nonseasonal MDD will be randomized into three groups (i.e. blue light, bright light or dim light). The treatment will be performed five times a week for the first two weeks. And for the next 2 weeks, the treatment for patients will be undertook three times a week. There will be 16 times in total. The investigators will assess nonseasonal MDD'symptom severity in the baseline, 1 week,2 week, 4 week,6 week and 8 week. Through the study, 17-item Hamilton Depression Rating Scale (HAMD17),14-item Hamilton Anxiety Rating Scale (HAMA14),Quick Inventory of Depressive Symptoms, Self-Rated version (QIDS-SR)，Pittsburgh sleep quality index (PSQI) , Clinical Global Impression scale(CGI), Quality of Life, Enjoyment and Satisfaction Questionnaire (Q-LES-Q),Morningness-Eveningness Questionnaire (MEQ),Repeatable Battery for the Assessment of Neuropsychological Status(RBANS),subjective fatigue symptom scale and semantic differential scale will be obtained. The patients will also get individual's data of heart rate and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for major depressive episodes as determined by MINI
* HAMD17≥17
* received antidepressive medication at stable dosages for at least 14 days

Exclusion Criteria:

* Any axis I psychiatric disorder comorbidity
* who have received formal psychological therapy, MECT or rTMS in 3 months
* any current significant medical condition especially eye diseases
* serious suicide risk
* pregnant or breastfeeding women
* depression with seasonal pattern
* treatment-resistant depression
* epilepsy in the past

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in 17-item Hamilton Depression Rating Scale (HAMD17) | from baseline to 8 weeks
  It assesses the severity of depression symptom. The responder on HAMD17 is defined as a HAMD17 decrease at least 50% from the baseline at post-treatment.

SECONDARY OUTCOMES:
Change in Quick Inventory of Depressive Symptoms, Self-Rated version (QIDS-SR) | from baseline to 8 weeks
  It's a self-rated inventory which assesses the severity of depression symptom
Change in 14-item Hamilton Anxiety Rating Scale (HAMA14) | from baseline to 8 weeks
  It assesses the severity of anxiety symptom.
Change in Pittsburgh sleep quality index (PSQI) | from baseline to 8 weeks
  It assesses the quality of sleep.
Change in Clinical Global Impression scale(CGI) | from baseline to 8 weeks
  It gives an overall clinical impression to the continuous outcome measures.
Change in Quality of Life, Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | from baseline to 8 weeks
  It assesses the quality of life, enjoyment and satisfaction
Change in Morningness-Eveningness Questionnaire (MEQ) | from baseline to 8 weeks
  It assesses the circadian phase
Change in Repeatable Battery for the Assessment of Neuropsychological Status(RBANS) | from baseline to 8 weeks
  It assesses cognitive function
Change in subjective fatigue symptom scale | from baseline to 8 weeks
  It assesses subjective fatigue symptom related to the light therapy
Change in semantic differential scale | from baseline to 8 weeks
  It assesses subjective feeling related to the light therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Wang, MD, Principal Investigator — Shanghai Zhongshan Hospital